CLINICAL TRIAL: NCT03958162
Title: The Comparison of Uniportal and Tubeless Video Assisted Thoracic Surgery and Transbronchial Lung Cryobiopsy Within the Multidisciplinary Discussion Context in the Diagnosis of Interstitial Lung Disease
Brief Title: The Comparison of Uniportal and Tubeless Video Assisted Thoracic Surgery and Transbronchial Lung Cryobiopsy in the Diagnosis of Interstitial Lung Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, ShiYue Li, Director of the Respiratory department, Guangzhou Institute of Respiratory Disease
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: TS20181008
Record Dates: First submitted 2019-05-20; First posted 2019-05-21 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Surgical Lung Biopsy; Transbronchial Lung Cryobiopsy; Interstitial Lung Disease
Keywords: surgical lung biopsy; transbronchial lung cryobiopsy; interstitial lung disease
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- uniportal and tubeless video assisted thoracic surgery (Experimental): lung biospy by the uniportal and tubeless video assisted thoracic surgery
  Interventions: Diagnostic Test: lung biopsy
- transbronchial lung cryobiopsy (Experimental): transbronchial lung cryobiopsy
  Interventions: Diagnostic Test: lung biopsy

INTERVENTIONS:
Diagnostic Test: lung biopsy — transbronchial lung cryobiopsy

SUMMARY:
To compariing the uniportal and tubeless video assisted thoracic surgery and trnsbronchial lung cryobiopsy within the multidisciplinary discussion context in the diagnosis of interstitial lung disease，and assess the safety and cost-effectiveness. This is a prospective control trial.

ELIGIBILITY:
Inclusion Criteria:

1. 18 yrs ≤ age<75yrs
2. Patients diagnosed as interstitial lung disease with comprehensive clinical data (including history, serological test, spirometry test and high resolution computed tomography)
3. Further pathological data was still required after multidisciplinary discussion.

Exclusion Criteria:

1. Severe pulmonary dysfunction: forced vital capacity (FVC) ≤65% or carbon-monoxide diffusion coefficient (DLco) ≤45% of predicted value
2. Pulmonary hypertension: An estimated systolic pulmonary artery pressure>50mmHg on echocardiography
3. Abnormal coagulation parameters or thrombocytopenia (<50*109/L)
4. Severe comorbidities leading to inoperable condition
5. Patients cannot give consent or refuse biopsy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Diagnotic yield | two weeks
  Percentage of definitive diagnosis within the multidisciplinary discussion context by two different biopsy methods

IPD SHARING:
Plan to Share IPD: Undecided